CLINICAL TRIAL: NCT02631746
Title: Phase II Trial of Nivolumab for HTLV-Associated Adult T Cell Leukemia/Lymphoma
Brief Title: Nivolumab in Treating Patients With HTLV-Associated T-Cell Leukemia/Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-02126; NCI-2015-02126 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 125462; 9925 (Other: Duke University - Duke Cancer Institute LAO); 9925 (Other: CTEP); UM1CA186704 (NIH)
Record Dates: First submitted 2015-12-15; First posted 2015-12-16 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Acute Adult T-Cell Leukemia/Lymphoma; Adult T-Cell Leukemia/Lymphoma; Chronic Adult T-Cell Leukemia/Lymphoma; HTLV-1 Infection; Lymphomatous Adult T-Cell Leukemia/Lymphoma; Smoldering Adult T-Cell Leukemia/Lymphoma
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; HTLV-I Infections | interventions — Nivolumab; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1. Treatment repeats every 14 days for 46 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacogenomic Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC

SUMMARY:
This phase II trial studies how well nivolumab works in treating patients with human T-cell leukemia virus (HTLV)-associated T-cell leukemia/lymphoma. Nivolumab is an antibody, which is a type of blood protein that tags infected cells and other harmful agents. Nivolumab works against a protein called programmed cell death (PD)-1 and may help the body destroy cancer cells by helping the immune system to keep fighting cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of nivolumab for patients with HTLV-associated adult T-cell leukemia lymphoma (ATLL).

II. To determine the efficacy of nivolumab for patients with HTLV-associated ATLL.

SECONDARY OBJECTIVES:

I. To determine effects of nivolumab on HTLV-1 proviral deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) loads.

II. To determine the effects of nivolumab on anti-HTLV-1 and anti-ATLL immune responses.

III. To determine effects of nivolumab on HTLV-1 integration site clonality.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 60 minutes on day 1. Treatment repeats every 14 days for 46 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any stage of pathologically confirmed cluster of differentiation (CD)3+ acute, lymphoma, chronic, or smoldering subtypes of ATLL
* Documentation of HTLV infection (enzyme linked immunosorbent assay [ELISA]) in individual with confirmation of HTLV-1 infection (by immunoblot or polymerase chain reaction [PCR]) or a consistent clinical picture (including two of the following: 1) CD4+ leukemia or lymphoma, 2) hypercalcemia, and/or 3) Japanese, Caribbean or South American birthplace)
* Patients with acute or lymphoma forms must have received at least one cycle of combination chemotherapy (with or without mogamulizumab) or interferon (with or without zidovudine and/or arsenic); individuals with chronic or smoldering acute T-cell lymphoma (ATL) are not required to have had prior treatment or could have received any number of previous courses of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky >= 60%)
* Life expectancy > 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation; women should continue birth control for 23 weeks after stopping nivolumab, and men should continue birth control for 31 weeks after stopping nivolumab; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 31 weeks after completion of nivolumab administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab
* Prior allogeneic transplantation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any condition requiring > 10 mg/d prednisone equivalents
* Current or prior HTLV-1 associated inflammatory diseases, including but not limited to myelopathy, uveitis, arthropathy, pneumonitis, or a Sjogren's disease-like disorder
* Prior treatment with anti-PD-1, anti-programmed death-ligand (PD-L)1, anti-PD-L2 antibody
* Grade 2 or greater toxicity from prior therapy
* Grade 2 or greater diarrhea
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies (other than HTLV-associated arthropathy), and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible; patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* Patients who have hepatitis C (both reactive anti-hepatitis C virus [HCV] antibody and detectable HCV RNA) and hepatitis B (hepatitis B surface antigen [HBsAg] positive and anti-hepatitis B core [HBc]-total positive), may be enrolled, provided their total bilirubin: =< 1.5 x institutional upper limit of normal (ULN) AST (SGOT)/ALT (SGPT): =< 2.5 x institutional upper limit of normal
* Patients with concurrent human immunodeficiency virus (HIV) infection may be enrolled if compliant with 3 or more drug anti-retroviral regimen and virus load less than 50 copies/ml and CD4 count greater than 250 cells/ml, and no concurrent opportunistic infection or other malignancy
* Any other prior malignancy from which the patient has been disease free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site or any other cancer
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, Principal Investigator — Duke University - Duke Cancer Institute LAO
Locations (6):
- United States (6):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Rauch DA, Conlon KC, Janakiram M, Brammer JE, Harding JC, Ye BH, Zang X, Ren X, Olson S, Cheng X, Miljkovic MD, Sundaramoorthi H, Joseph A, Skidmore ZL, Griffith O, Griffith M, Waldmann TA, Ratner L. Rapid progression of adult T-cell leukemia/lymphoma as tumor-infiltrating Tregs after PD-1 blockade. Blood. 2019 Oct 24;134(17):1406-1414. doi: 10.1182/blood.2019002038. PMID 31467059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 3
Completed | 0
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events of Nivolumab, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicity by grade will be summarized using descriptive statistics. The incidence of toxicities will be estimated using the binomial proportion and its 90% confidence interval.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Tumor Response, Evaluated Using the New International Criteria Proposed by the Revised Response Evaluation Criteria in Solid Tumors Guideline (Version 1.1)
Description: Summarized using descriptive statistics. Binomial proportions and their 90% confidence intervals will be used to estimate the response rates of therapy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Duration of Response
Description: Summarized using descriptive statistics. Binomial proportions and their 90% confidence intervals will be used to estimate the response rates of therapy. The Kaplan-Meier method will be used to evaluate the response duration.
Time Frame: 1 year
Population: Duration of response cannot be calculated because of no responders.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Effects of Treatment
Description: Analysis of variance methods will be used to evaluate the effects of treatment.
Time Frame: 1 year
Population: Post-treatment data not available because no patients made it to Cycle 3 Day 1.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Time on the Viral Load Measurements
Description: Analysis of variance methods will be used to evaluate the effects of treatment and time on the viral load measurements, as well as measurements of viral transcripts. A proportional hazards analysis with viral load measures as time dependent covariates will be used to evaluate the effects of these measures on duration of response.
Time Frame: 1 year
Population: Post-treatment data not available because no patients made it to Cycle 3 Day 1.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

6. Secondary Outcome: HTLV-1 Clonality
Description: Measured from peripheral blood mononuclear cell (PBMC) samples.
Time Frame: 1 year
Population: Post-treatment data not available because no patients made it to Cycle 3 Day 1.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

7. Secondary Outcome: HTLV-1 Specific Cytotoxic T Lymphocytes (CTLs)
Description: Measured from PBMC samples.
Time Frame: 1 year
Population: Post-treatment data not available because no patients made it to Cycle 3 Day 1.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

8. Secondary Outcome: Immune Cell Numbers
Description: Measured from blood and tissue samples.
Time Frame: 1 year
Population: Post-treatment data not available because no patients made it to Cycle 3 Day 1.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=3)
Abdominal Pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Splenomegaly/splenic infarct (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=3)
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Blood bilirubin increased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Creatinine increased (Investigations) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
INR increased (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT02631746/Prot_SAP_000.pdf